CLINICAL TRIAL: NCT03602729
Title: Comparison of Teaching Interventions to Improve Breastfeeding Among Mothers of Infants In Neonatal Intensive Care Unit of Brookdale Hospital Medical Center
Brief Title: Comparison of Breastfeeding Teaching Intervention
Acronym: BFTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brookdale University Hospital Medical Center (Other)
Responsible Party: Principal Investigator, Surichhya Bajracharya, Resident in pediatrics, Brookdale University Hospital Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18-02
Record Dates: First submitted 2018-05-30; First posted 2018-07-27 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Breast Feeding
Keywords: Breastfeeding; Teaching; Intervention; NICU
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (No Intervention): No study related education given
- Group 2 (Experimental): Written BF education
  Interventions: Other: Breastfeeding education
- Group 3 (Experimental): Verbal BF education
  Interventions: Other: Breastfeeding education
- Group 4 (Experimental): Video BF education
  Interventions: Other: Breastfeeding education

INTERVENTIONS:
Other: Breastfeeding education — Breastfeeding education in three different forms: written/verbal/video
  Arms: Group 2; Group 3; Group 4

SUMMARY:
Investigators plan to include mother-infant couplets admitted to Neonatal Intensive Care Unit(NICU) at Brookdale Hospital for clinical reasons during one year period 1/2018-1/2019. Participants whose infants have health conditions that will not allow breastfeeding, not able to read or understand English and/or participants refusing to provide phone numbers, an email address or mail address for future communication will not be included in the study.

After obtaining an informed consent, participants will be allocated to one of the four study groups by randomization and participants will receive either no education or one of the verbal/written/video education at two different time points: within 4 days and at 2 weeks from the time of birth of the infant. Participants whose infants are in NICU and are feeding expressed breastmilk will be instructed to bring all the expressed breastmilk to NICU and to keep records of the date, time and the amount of expressed breastmilk in the log book maintained at the bedside of the infant. Participants who are directly feeding the infant on breast will be contacted by third personnel who is blind to which study group the participant belongs to qualitatively evaluate breast feeding in terms of frequency, duration, exclusive breast feeding at 2 weeks, 4 weeks and 6 weeks from the time of birth. Participants will be requested not to reveal the study team about the mode of teaching method she has received when she is contacted at 2 weeks, 4 weeks and 6 weeks for the evaluation of the breast feeding. Investigators will also go through the medical records of participants and their infants to collect some demographic data and clinical characteristics pertinent for the study such as age, parity, weight of the infant.

Thus, investigators plan to compare the breast-feeding outcome quantitatively among participants who are feeding expressed breast milk and qualitatively as duration/exclusive breast-feeding among participants who are feeding directly on breast following three different teaching interventions: written or verbal or video and find out the most effective method of teaching intervention

DETAILED DESCRIPTION:
The purpose of the study is to compare the breast-feeding outcome following three different teaching interventions: written or verbal/direct or visual/videos among participants whose infants are admitted in Neonatal Intensive Care Unit (NICU) at Brookdale Hospital

1. Breast-feeding outcome among participants who are feeding expressed breast milk will be measured quantitatively as amount of milk production per day on an average during NICU stay.
2. Breast-feeding outcome among participants who are directly feeding the infants at breast will be measured qualitatively in terms of frequency, duration, exclusive breast feeding at 2 weeks, 4 weeks and 6 weeks of infant's life.

CLINICAL SIGNIFICANCE Investigators are including participants whose infants are admitted to the Brookdale NICU This also include very preterm [<32 weeks] infants, the period when breastfeeding incidence has been lesser compared to participants who give birth at later gestation and those who don't require admission to NICU. By including participants who give birth <32 weeks and newborns admitted to NICU, investigators will be able to document the quantity of breast milk production by logging the milk brought to our NICU storage freezer by participants and effectively measure the outcome objectively of the three different interventions [written, verbal and visual methods].

Previous studies have found that breast feeding is lower among African American population. Since most of population at Brookdale hospital is African American, this study will also give an opportunity to find the result of education intervention among this population Investigators propose that this study will be useful to find the most effective mode to educate participants whose neonates admitted to NICU about breast-feeding and may enhance the culture of breastmilk feeding in this population and therefore increase breast feeding among newborns admitted to the NICU.

METHODOLOGY This is a prospective randomized study on breast-feeding teaching intervention on participants who give birth to newborns that are admitted to NICU at Brookdale Hospital during one-year period 1/2018-1/2019.

All participants who deliver at Brookdale hospital receive regular breast-feeding education on benefit of exclusive breastfeeding, latching, pumping provided by the nurses or physicians during postpartum period while they are admitted in the hospital. The participants also receive education on breastfeeding through public health assistant/volunteer through New York City (NYC) Family and Child Health Bureau of Maternal Infant and Reproductive Health either at the hospital and or during home visit following discharge.

Any education provided as a part of research is the additional education participant will receive on top of the regular education all participants receive irrespective of their participation and the group they belong to in the study. Participant decision to participate or not in the study will not affect the regular health care and education participant or participant's infant will receive in the hospital.

The aim of the study is to obtain at-least 25 participants per group for a total sample size of 100 participants and 100 participants' infants.

Once investigators identify the participants fulfilling the inclusion criteria, one of the two trained investigators will take an informed consent that include permission to contact participants over the phone or by email/mail at 2 weeks, 4 weeks and 6 weeks for providing the appropriate method of teaching intervention and/ or measurement of breast feeding outcome.

Randomization will be done by picking up one of the random numbers representing each group such as 1 for Group 1, 2 for Group 2, 3 for Group 3 and 4 for Group 4:

Group 1: Participants in this group will not receive additional teaching interventions included in the research. Participants will be contacted at 2 weeks, 4 weeks and 6 weeks postpartum to evaluate amount, duration, exclusive breast feeding.

Group 2: Participants in this group will receive the written breast-feeding education in the form of booklet (included with this protocol). Booklet will be distributed 2 times: 1st time in the hospital within 4 days of birth of the infant before the participant is discharged and at 2 weeks from the time of birth of the infant utilizing the time when participant visits to the NICU. If the participant is not able to visit NICU or the infant is discharged from the hospital before 2 weeks from the time of birth, booklet will be provided to the participant by post or as an attachment in an email. Participants will be contacted at 2 weeks, 4 weeks and 6 weeks postpartum to evaluate amount, duration, exclusive breast feeding Group 3: Participants in this group will receive breast-feeding education verbally (please find the content of verbal education in following page). Verbal education will be provided 2 times: 1st time in the hospital within 4 days of birth of the infant before the participant is discharged. Subsequent breast-feeding trouble shooting verbal education will be provided at 2 weeks from the time of birth of the infant utilizing the time when participant visits to the NICU. If the participant is not able to visit NICU or the infant is discharged from the hospital before 2 weeks from the time of birth, verbal education will be provided to the participant over the phone. Participants will be contacted at 2 weeks, 4 weeks and 6 weeks postpartum to evaluate amount, duration, exclusive breast feeding Group 4: Participants in this group will receive breast-feeding education through the video format. (links for the video is provided in the following page). Video education will be provided 2 times: 1st time in the hospital within 4 days of birth of the infant before the participant is discharged. Subsequent breast-feeding video education will be provided at 2 weeks from the time of birth of the infant by sending a link for the video in participant's email. Participants will be contacted at 2 weeks, 4 weeks and 6 weeks postpartum to evaluate amount, duration, exclusive breast feeding All three forms of education will include similar information that include advantages of breast-feeding, optimization of pumping using hand pump or electric pump, storage of milk and such other troubleshooting during breastfeeding

Written education method:

Written education will be provided in the form of booklet. Investigators have received 100 booklets 'your guide to breastfeeding' from The U.S. Department of Health and Human Services Office on Women's Health (OWH) for free. Investigators will provide the booklet to the participants that belong to group 2 as written education within 4 days of the birth of the infant and at 2 weeks from the time of birth of the infant.

This standard booklet can be found free at the government website below: https://www.womenshealth.gov/files/documents/your-guide-to-breastfeeding.pdf

Verbal education method:

Verbal education will be provided by one of the two investigators who will use the checklist to provide the information. Both investigators have successfully completed online "Supporting and Promoting Breastfeeding in Health Care Settings modules' from School of Public Health, University of Albany, State University of New York. Both investigators will be trained by a neonatologist so that the verbal education method provided by two different investigators is similar. The checklist in verbal education is derived from the above standard booklet so that the information provided is same as the booklet.

Video education method:

There is standard you-tube video link for free at the following government website:

https://www.womenshealth.gov/printables-and-shareables/resource/videos Participants will be provided you-tube video links included in the following table within 4 days and at 2 weeks from the time of birth of the infant.

ELIGIBILITY:
Inclusion Criteria:

* Mother-infant couplets with newborns admitted to NICU at Brookdale Hospital for clinical reasons.

Exclusion Criteria:

* Any contraindications to breast-feeding such as galactosemia, protein milk allergy, HIV infection, maternal substance abuse
* Mothers not able to read and/or understand English
* Mothers refusing to provide phone number or an email address or mail address for future communication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
amount of breast milk expression | 2 weeks
  amount of breast milk expression in milliliters
Duration of breast feeding | 2 weeks
  Duration of breast feeding in weeks
Frequency of breast feeding | 2 weeks
  Frequency of breast feeding in number of times in a day
Exclusive breast feeding | 2 weeks
  Exclusive breast feeding as yes or no
amount of breast milk expression | 4 weeks
  amount of breast milk expression in milliliters
amount of breast milk expression | 6 weeks
  amount of breast milk expression in milliliters
Duration of breast feeding | 4 weeks
  Duration of breast feeding in weeks
Duration of breast feeding | 6 weeks
  Duration of breast feeding in weeks
Frequency of breast feeding | 4 weeks
  Frequency of breast feeding in number of times in a day
Frequency of breast feeding | 6 weeks
  Frequency of breast feeding in number of times in a day
Exclusive breast feeding | 4 weeks
  Exclusive breast feeding as yes or no
Exclusive breast feeding | 6 weeks
  Exclusive breast feeding as yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Surichhya Bajracharya, Principal Investigator — Brookdale University Hospital Medical Center; Sravanti Kurada, Study Director — Brookdale University Hospital Medical Center
Locations (1):
- Brookdale University hospital and Medical Center, Brooklyn, New York, United States